CLINICAL TRIAL: NCT00430378
Title: Acupuncture for Prevention of Radiation-Induced Xerostomia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2006-0763; NCI-2012-02115 (Registry Identifier: NCI CTRP); U19CA121503 (NIH)
Record Dates: First submitted 2007-01-30; First posted 2007-02-01 (Estimated); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Xerostomia; Mouth Dryness; Nasopharyngeal Cancer
Keywords: Xerostomia; Dry Mouth; Mouth Dryness; Nasopharyngeal Cancer; Acupuncture
MeSH Terms: conditions — Xerostomia; Nasopharyngeal Neoplasms | interventions — Acupuncture Therapy; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture (Experimental): Acupuncture Before the Radiation Treatment
  Interventions: Procedure: Acupuncture
- Standard Care (Experimental): Standard Care Without Acupuncture
  Interventions: Other: Standard Care

INTERVENTIONS:
Procedure: Acupuncture — Acupuncture for 20 minutes before the radiation therapy session, 3 days a week for 7 weeks.
  Arms: Acupuncture
Other: Standard Care — No Acupuncture.
  Arms: Standard Care

SUMMARY:
The goal of this clinical research study is to learn if acupuncture is effective in preventing xerostomia (dry mouth) in cancer patients who receive radiation treatment to the head and neck area. Researchers also want to learn whether acupuncture lowers the severity of dry mouth that is experienced by these patients.

Primary Objective:

-Investigate if acupuncture is effective in preventing xerostomia among cancer patients at Fudan University Cancer Hospital (Cancer Hospital) who receive radiation treatment to the head and neck area.

Secondary Objectives:

* Determine whether acupuncture reduces the severity of xerostomia.
* Determine the feasibility of providing acupuncture treatment to patients at Cancer Hospital who are receiving radiation treatment for cancer of the head and/or neck area.

DETAILED DESCRIPTION:
Some research suggests that acupuncture may be helpful in stimulating saliva flow in patients with dry mouth caused by radiation treatment. Acupuncture uses very thin needles inserted at certain points on the body that are believed to affect bodily functions.

Before you can start treatment on this study, you will have "screening tests." These tests will help the doctor decide if you are eligible to take part in this study. Your complete medical history will be recorded, and you will have a physical exam. You will also be asked to complete 3 short questionnaires about your quality-of-life and current saliva flow. These should take about 5 minutes to complete. You will be asked to collect saliva in a vial (small tube or jar) for 5 minutes, by allowing saliva to collect in your mouth and then spitting it into the vial. You will be asked to collect saliva twice at each time point. One collection will be like it is described above. The second collection will be after you have held a sour liquid in your mouth for 1 minute. A traditional Chinese medicine diagnosis will also be conducted. This will include diagnosis by a doctor as well as by using a heart-rate machine and taking a photograph of your tongue. This will allow a more objective check of your heart rate and tongue condition.

If you are found to be eligible to take part in the study, you will be randomly assigned (as in the toss of a coin) into 1 of 2 groups. One group will receive acupuncture during their radiation treatment period, and the other will receive standard care without acupuncture. Participants assigned to the acupuncture group will receive acupuncture for 20 minutes before their radiation therapy session, 3 days a week for 7 weeks. Participants in the standard care group will not receive acupuncture.

If you are in the acupuncture group, you will be asked to come to the acupuncture clinic for the treatment, before your radiation treatment. The acupuncturist will put in the needles in certain points of your body (including the chin, wrist, leg, and ear), while you are seated in a chair. The needles will remain in for about 20 minutes.

If you choose to receive medications for dry mouth at any point while on study, your participation on this study will end.

No matter which group you are assigned to, for each of the 7 weeks you are receiving radiation treatment, your vital signs (your blood pressure and pulse) will be checked, and you will be asked about any medications you are taking. You will also complete questionnaires about your quality-of-life and symptoms. Each questionnaire should take about 5 minutes to complete. A saliva sample will also be collected on Weeks 1, 3, 4, 6, and 7. If you are assigned to the acupuncture group, the saliva sample will be collected after the acupuncture treatment on Weeks 1, 4, and 7 and before the treatment on Weeks 3 and 6. A traditional Chinese medicine diagnosis will also be conducted in the middle of radiation treatment, at the end of treatment, and 1 month later. This will include diagnosis by a physician as well as by using a pulse machine and taking a photograph of your tongue.

One month after the end of radiation treatment (Week 11), your vital signs will be checked, you will be asked about any medications you are taking， you will complete the quality of life and symptom questionnaires, and you will provide another saliva sample. After Week 11, your participation on this study is over.

This is an investigational study. Up to 100 patients will take part in this study. All will be enrolled at the Fudan University Cancer Hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Adult >/= 18 year of age and able to sign informed consent
2. Diagnosed with nasopharyngeal carcinoma and scheduled to undergo concurrent chemotherapy and radiation treatment
3. Treatment plan must include treatment of at least 50 gray bilateral to the parotid
4. Must have anatomically intact parotid and submandibular glands
5. Karnofsky Performance Status > 60
6. If the participant is female and of child bearing potential, must have a negative urine pregnancy test.

Exclusion Criteria:

1. History of xerostomia prior to the head and neck radiation therapy (Sjögren's disease or other underlying systemic illness known to cause xerostomia).
2. Planned IMRT
3. Suspected or confirmed physical closure of salivary gland ducts on either side
4. Known bleeding disorders and on Heparin or Coumadin
5. Upper or lower extremity deformities that could interfere with accurate acupoint location or alter the energy pathway as defined by traditional acupuncture theory
6. Local skin infections at or near the acupuncture site or active systemic infection
7. History of cerebrovascular accident or spinal cord injury. (The mechanism of action for acupuncture may be associated with central nervous system (CNS) activity, and patients with CNS pathology may respond differently to treatment than the general population.)
8. Mental incapacitation or significant emotional or psychiatric disorder that, in the opinion of the investigator, precludes study entry as these patients may not be able to cooperate with this slightly invasive procedure or with the data collection process
9. Current acknowledged use of any illicit drugs or evidence of alcohol abuse as defined by The American Psychiatric Association criteria
10. Participants who are taking or who have taken any investigational new drug within the last 30 days, or who are planning to take such a drug during the course of the study
11. Current acknowledged use of other alternative medicines such as herbal preparations that could affect salivary function. Each patient will be asked for a list of herbal supplements they are currently taking and this will be reviewed on an individual basis. Patients will be excluded if they are taking any herbs known or suspected to affect salivary function
12. Participants taking cholinergic agonist medication (Pilocarpine, Cevimeline), beta adrenergic antagonists, anticholinergic agents or other medications known to affect salivary function
13. Currently receiving acupuncture for any condition
14. No prior head and neck radiation treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-01 (Actual); Primary Completion 2021-05-27 (Actual); Study Completion 2021-05-27 (Actual)

PRIMARY OUTCOMES:
Number of Patients with Xerostomia | Baseline + 8 additional points in time (baseline, weeks1-7, week 11).
  Severity of the xerostomia in both groups compared by testing for group differences in xerostomia scores between baseline and week 7 using a two-sample (unpaired) t test. Repeated measures analyses used in order to detect overall differences in severity over time, differences between groups and the interaction between time and group.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph S. Chiang, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- Fudan University Cancer Hospital, Shanghai, China

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org